CLINICAL TRIAL: NCT00507117
Title: Prospective, Randomized, Placebo Controlled Trial Assessing the Effects of Ezopiclone on the Quality of Overnight Polysomnography and CPAP Titration
Brief Title: Ezopiclone Improves the Quality of Overnight Polysomnography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: WRAMC05-17017
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Polysomnography; Non-benzodiazepine hypnotics
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Eszopiclone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PSG (Active Comparator)
  Interventions: Drug: Lunesta; Drug: Placebo control

INTERVENTIONS:
Drug: Lunesta — Lunesta 3mg prior to PSG
Drug: Placebo control — matching placebo

SUMMARY:
Patients often have difficulty sleeping during overnight sleep testing in a lab environment. The purpose of this study is to determine if taking a sleep aid will improve sleep and therefore the quality of the sleep study.

DETAILED DESCRIPTION:
The increasing awareness of sleep-disordered breathing (i.e obstructive sleep apnea) has created a growing demand for polysomnography (sleep study), resulting in excessive waiting times in many laboratories. Sleep centers have therefore needed to develop methods to improve their efficiency. Unfortunately many patients find it difficult to fall asleep in the unfamiliar environment of a laboratory setting (the "first-night effect"), circumstances that may prolong falling alseep and staying sleep. Likewise, intolerance of continuous positive airway pressure (CPAP) may also reduce the quality of the sleep study. Poor quality studies may lead to an inability to make a diagnosis or adequately titrate CPAP therapy. Unsatisfactory studies may need to be repeated.

Sleep aids (hypnotics) are commonly used to treat both acute and chronic insomnia. These agents have minimal side-effects and do not disrupt normal sleep architecture or alter respiratory events. These attributes make such agents ideal for use to improve the quality of sleep studies and enhance the efficiency of sleep centers.

In a recent retrospective review, we found that the use of a hypnotic prior to the sleep study resulted improved patient satisfaction and improved quality of the sleep study with significantly less studies needing to be repeated. Although promising, these results must be validated with a prospective, randomized, placebo-controlled trial.

Eszopiclone (Lunesta) is a new non-narcotic, non-benzodiazepine hypnotic agent which received FDA approval on December 15, 2004 for the treatment of acute and chronic insomnia. Multiple clinical trials have found that eszopiclone decreases sleep latency, improves sleep efficiency/maintenance and reduces wake time after sleep onset (WASO). Given its efficacy in promoting sleep onset and sleep maintenance and its excellent safety profile, this agent should be ideal as a pre-study sedative. The purpose of this study is to validate the use of Lunesta in improving the quality of overnight sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients aged 18-65, evaluated by a sleep medicine provider in the Walter Reed Army Medical Center Sleep Disorders Clinic, who are referred for PSG for suspected Obstructive Sleep Apnea Syndrome

Exclusion Criteria:

* Pregnancy
* Liver dysfunction or history of EtOH abuse
* Concomitant use of benzodiazepines, narcotics or ketozonazole
* Decompensated CHF
* CVA within 3 months
* Uncontrolled psychiatric disorders
* Patients < 18 years old
* Patients over 65

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
diagnostic yield of PSG | during overnight study
total sleep time | during overnight study
wake after sleep onset | during overnight study
sleep latency | during overnight study
sleep efficiency | during overnight study
total arousal index | during overnight study
respiratory disturbance index at highest CPAP level | during overnight study

SECONDARY OUTCOMES:
Respiratory Disturbance Index | during overnight study

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Lettieri, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Lettieri CJ, Eliasson AH, Andrada T, Khramtsov A, Kristo DA. Does zolpidem enhance the yield of polysomnography? J Clin Sleep Med. 2005 Apr 15;1(2):129-31. PMID 17561625
- [Derived] Lettieri CJ, Collen JF, Eliasson AH, Quast TM. Sedative use during continuous positive airway pressure titration improves subsequent compliance: a randomized, double-blind, placebo-controlled trial. Chest. 2009 Nov;136(5):1263-1268. doi: 10.1378/chest.09-0811. Epub 2009 Jun 30. PMID 19567493
- [Derived] Lettieri CJ, Quast TN, Eliasson AH, Andrada T. Eszopiclone improves overnight polysomnography and continuous positive airway pressure titration: a prospective, randomized, placebo-controlled trial. Sleep. 2008 Sep;31(9):1310-6. PMID 18788656